CLINICAL TRIAL: NCT03895697
Title: A Phase 3b, Randomized, Double-blind, Crossover Trial to Compare the Efficacy and Safety of 2 Different Batches of Subcutaneous Dasiglucagon in Patients With Type 1 Diabetes Mellitus
Brief Title: A Trial to Compare the Efficacy and Safety of 2 Different Batches of Subcutaneous Dasiglucagon in Patients With T1DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-17084
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
Keywords: glucagon
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — dasiglucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dasiglucagon batch A crossover to dasiglucagon batch B (Experimental): V2: Single fixed dose (subcutaneous injection) of dasiglucagon batch A then at V3: Single fixed dose (subcutaneous injection) of dasiglucagon batch B
  Interventions: Drug: dasiglucagon
- Dasiglucagon batch B crossover to dasiglucagon batch A (Experimental): V2: Single fixed dose (subcutaneous injection) of dasiglucagon batch B then at V3: Single fixed dose (subcutaneous injection) of dasiglucagon batch A
  Interventions: Drug: dasiglucagon

INTERVENTIONS:
Drug: dasiglucagon — Glucagon analogue
  Other Names: ZP4207

SUMMARY:
A randomized, double-blind, crossover trial to compare the efficacy and safety of 2 different batches of subcutaneous dasiglucagon in patients with type 1 diabetes mellitus (T1DM)

DETAILED DESCRIPTION:
This multicenter, double-blind, crossover, randomized clinical trial was designed to evaluate the efficacy and safety of 2 different batches of subcutaneous dasiglucagon in patients with T1DM. Patients were randomly assigned 1:1 to either dasiglucagon Batch A or dasiglucagon Batch B as their initial dose and the other as the second dose. To avoid bias in the evaluation of clinical assessments, the trial was conducted in a double-blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 1 year according to the diagnostic criteria as defined by the American Diabetes Association.
* Hemoglobin A1c <10.0% at screening
* Treated with stable insulin treatment (defined as no more than a 10-unit daily variation in total daily insulin dose) 30 days prior to screening

Exclusion Criteria:

* History of hypoglycemic events associated with seizures in the last year prior to screening
* History of severe hypoglycemia (an episode requiring assistance from another person) in the last month prior to screening
* Previous participation in a clinical trial within the dasiglucagon program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Time to plasma glucose recovery | 0-45 minutes after dosing
  Plasma glucose recovery is defined as first increase in plasma glucose of ≥20 mg/dL (1.1 mmol/L) from baseline during the hypoglycemic clamp procedure without administration of rescue intravenous glucose

SECONDARY OUTCOMES:
Plasma glucose changes from baseline | 0-30 minutes after dosing
  Plasma glucose changes from baseline at 30 minutes, at 20 minutes, at 15 minutes, and at 10 minutes after trial drug injection or at the time of rescue patient level).
Pharmacodynamics - Area under the effect curve 30 min | 0-30 minutes after dosing
  Area under the baseline-adjusted effect curve (AUE) from zero up to the concentration at 30 minutes, AUE 0-30min
Pharmacodynamics - Area under the effect curve 90 min | 0-90 minutes after dosing
  Area under the baseline-adjusted effect curve (AUE) from zero up to the concentration at 90 minutes, AUE 0-90min
Pharmacodynamics - Maximum plasma glucose concentration | 0-90 minutes after dosing
  Change from baseline plasma glucose to maximum plasma glucose measure after dosing, CEmax
Pharmacodynamics - Time maximum plasma glucose concentration | 0-90 minutes after dosing
  Time to maximum change in plasma glucose measure from baseline, TEmax
Pharmacokinetics - Area under the plasma concentration-time curve 30 min | 0-30 minutes after dosing
  Area under the concentration-time curve (AUC) from zero up to the concentration at 30 minutes, AUC0-30min
Pharmacokinetics - Area under the plasma concentration-time curve 300 min | 0-300 minutes after dosing
  Area under the concentration-time curve (AUC) from zero up to the concentration at 300 minutes, AUC0-300min
Pharmacokinetics - Area under the plasma concentration curve Infinitely | 0-300 minutes after dosing
  Area under the concentration-time curve from zero up to the concentration at infinitely after dosing, AUC0-inf
Pharmacokinetics - Maximum plasma concentration | 0-300 minutes after dosing
  Measured maximum plasma drug concentration after dosing, Cmax
Pharmacokinetics - Time to maximum plasma concentration | 0-300 minutes after dosing
  Sampling time until reaching Cmax, Tmax
Pharmacokinetics - Half-life | 0-300 minutes after dosing
  Half-life dasiglucagon, t½
Pharmacokinetics - Volume of distribution | 0-300 minutes after dosing
  Apparent volume of distribution of dasiglucagon, Vz/f
Pharmacokinetics - Mean residence time | 0-300 minutes after dosing
  Mean residence time, MRT
Pharmacokinetics - Body clearance | 0-300 minutes after dosing
  Total body clearance, CL/f
Safety - Adverse events | 90 days
  The incidence, type and severity of adverse events (AEs)
Safety - Number of rescue infusions | 0-90 minutes after dosing
  Number of rescue infusions of IV glucose after trial drug administration
Safety - Time to first rescue infusion | 0-90 minutes after dosing
  Time to first rescue infusion of IV glucose after trial drug administration
Immunogenicity - Occurrence of anti-drug antibodies | 60 days
  Occurrence of antibodies against dasiglucagon

CONTACTS AND LOCATIONS:
Overall Officials: Stine J Maarbjerg, PHD, Study Director — Zealand Pharma A/S
Locations (1):
- LMC Diabetes & Manna Research, Toronto, Ontario, Canada